CLINICAL TRIAL: NCT02651207
Title: Study Looking at Acceptability of Using Ethyl Chloride Spray Versus Subcutaneous Lidocaine Anaesthetic Prior to Contraceptive Implant Insertion
Brief Title: Ethyl Chloride Spray Versus Subcutaneous Lidocaine Anaesthetic Prior to Contraceptive Implant Insertion
Status: Withdrawn | Type: Observational
Why Stopped: decided not to do study. This will be run as a service evaluation instead
Sponsor: Tayside Medical Science Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 2015OB09
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- local anaesthetic spray group: women will either chose the above, ethyl chloride spray prior to having their contraceptive implant fitted or the below injection. This comes in a canister and a maximum of 5 spray for 5 seconds will be applied topically to the skin at the site of the contraceptive implant insertion
  Interventions: Other: Questionnaire based study looking at pain scores felt by patients either having a lidocaine injection or ethyl chloride spray prior to insertion of a contraceptive implant
- local anaesthetic injection group: women will either chose ethyl chloride spray prior to having their contraceptive implant fitted or the injection, subcutaneous 1% lidocaine, usually a dose of about 1-2 mls to the area skin where the contraceptive implant is to be inserted.
  Interventions: Other: Questionnaire based study looking at pain scores felt by patients either having a lidocaine injection or ethyl chloride spray prior to insertion of a contraceptive implant

INTERVENTIONS:
Other: Questionnaire based study looking at pain scores felt by patients either having a lidocaine injection or ethyl chloride spray prior to insertion of a contraceptive implant

SUMMARY:
Study to look at the acceptability of local anaesthetic spray versus injection, prior to contraceptive implant insertion

DETAILED DESCRIPTION:
Currently, patients undergoing contraceptive implant insertion are offered local anaesthetic with an injection before insertion. This study aims to look at whether patients find using the local anaesthetic spray more acceptable or equally acceptable to using local anaesthetic injection. Both are currently licensed products for use as skin anaesthesia but the spray is potentially quicker and involves less injections. Some areas of sexual health are already offering this option but there isn't much evidence as to which patients find more acceptable.

Patients in this study will be given a choice of anaesthetic asked to complete a short questionnaire, giving a pain score , on the pain rating scale of 0 to 10, ( being no pain to 10 being extremely painful. ) In addition, they will be asked to give the reasons for their choice. The questionnaire will be anonymous.

Average pain scores will be calculated between in group and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patient has chosen to use the implant as a method of contraception
* Patients will be assessed for medical eligibility for the contraceptive implant have no contraindications to either the implant, lidocaine or the ethyl chloride spray. However, if they have a known sensitivity to either the spray or the lidocaine ejection, they will be offered the other.
* Age between 13 and 55
* Has capacity to consent
* Has read the information sheet and consents to the study
* This will be offered for insertions of implant only i.e. not implant removals

Exclusion Criteria:

* Has a contraindication to have a contraceptive implant
* Doesn't wish to have a implant
* Allergy to either the implant, the lidocaine, the ethyl chloride or any of the incipient ingredients. Although patients will be given the option, if they have an allergy/contraindication to one of the products, they will be offered the other
* Is under 13 or over 55

Ages: 13 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patient who choose to use the contraceptive implant as a method of contraception and who are deemed medically eligible for the method with no medical contrainidications
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
acceptability of using ethyl chloride spray versus subcutaneous lidocaine anaesthetic prior to contraceptive implant insertion | one year
  Questionnaire based study looking at pain scores on the numeric pain rating scale 0 to 10, 0 being no pain to 10 being extremely painful

SECONDARY OUTCOMES:
acceptability of using ethyl chloride spray versus subcutaneous lidocaine anaesthetic prior to contraceptive implant insertion | one year
  Questionnaire looking at the reasons why women chose to use the injection or the spray

IPD SHARING:
Plan to Share IPD: No